CLINICAL TRIAL: NCT02471599
Title: Effect of Tonsillectomy on Longterm Renal Outcome of IgA Nephropathy :a Prospective,Randomized,Controlled Study.
Brief Title: Effect of Tonsillectomy on Longterm Renal Outcome of IgA Nephropathy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was suspended because that few participants was enrolled.
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGNSIgAN-003
Record Dates: First submitted 2015-05-19; First posted 2015-06-15 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; tonsillitis; tonsil provocation test; Tonsillectomy
MeSH Terms: conditions — Glomerulonephritis, IGA; Tonsillitis | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tonsillectomy group (Experimental): The case group will receive tonsillectomy.
  Interventions: Procedure: tonsillectomy
- non-tonsillectomy group (Active Comparator): The controlled group will not receive tonsillectomy.
  Interventions: Other: non-tonsillectomy

INTERVENTIONS:
Procedure: tonsillectomy — The tonsillectomy will be performed by the otolaryngologist. In addition, all subjects will receive the conventional drug treatments, defined as treatment of participants using the angiotensin-converting enzyme inhibitor (ACEi)/angiotensin II receptor blocker (ARB), anticoagulants, antihypertensives, corticosteroids so on, according to individual status.
  Arms: tonsillectomy group
Other: non-tonsillectomy — The non-tonsillectomy group received conventional drug treatments defined as treatment of participants using the ACEi/ARB,Anticoagulants, Antihypertensives, corticosteroids and so on, according to individual status.
  Arms: non-tonsillectomy group

SUMMARY:
The effect of tonsillectomy therapy on IgA nephropathy is still controversial.Few prospective,randomized investigations have examined how tonsillectomy affects the shortterm and longterm renal outcome of IgA nephropathy.This is A prospective,randomized ,controlled study to explore the longterm effect of tonsillectomy for patients with IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to sign an informed consent
* Age:18~45 years, regardless of gender
* Clinical evaluation and renal biopsy diagnostic for immunoglobulin A nephropathy (IgAN), excluded secondary IgAN. Renal histological criteria should be defined by Lee's glomerular grading system.
* Any one of three Tonsilar conditions defined by Otorhinolaryngologist : 1,recurrent acute tonsillitis accompanied with gross hematuria or urinary findings abnormality；2,recurrent acute tonsillitis without gross hematuria，but tonsil provocation test was positive；3, No history of acute tonsillitis,body examination found hypertrophy or atrophy tonsils ,crypt pus of tonsils ,or scars on the tonsil surface ,and positive tonsil provocation test.
* Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2

Exclusion Criteria:

* Inability or unwillingness to sign the informed consent
* Inability or unwillingness to meet the scheme demands raised by the investigators
* Rapidly progressive nephritic syndrome and acute renal failure, 24-hour urine protein≥3.5g,including rapidly progressive IgAN (IgAN with rapid decline in renal function characterized histologically by necrotizing vasculitis and crescent formation≥30%) necessitating the use of other immunosuppressive agents.
* Secondary IgAN such as systemic lupus erythematosus, Henoch-Schonlein purpuric nephritis and hepatitis B -associated nephritis
* est GFR < 30 mL/min/1.73m2
* Malignant hypertension that is difficult to be controlled by oral drugs
* Cirrhosis, chronic active liver disease.
* History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease.)
* Any Active systemic infection or history of serious infection within one month of entry or known infection with HIV, hepatitis B, or hepatitis C.
* Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure , chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases)
* Malignant tumors (except fully cured basal cell carcinoma)
* Current or recent (within 30 days) exposure to any other investigation
* Current exposure to mycophenolic mofetil (MMF),azathioprine or corticosteroids. In case of current treatment with oral steroid ,entry is permitted after corticosteroids dosage below 0.4mg/kg per day.
* Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception
* Tonsillectomy had been done when IgAN diagnosis or known contraindication to tonsillectomy(such as neutropenia，bleeding tendency，or anatomic abnormalities）

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Renal survival rate or Deterioration of renal function | Every 12months for 10 years after tonsillectomy
  Deterioration of renal function (evidenced by a 50% rise from baseline serum creatinine (SCr) levels, or a 25% decline from baseline estimated glomerular filtration rate (eGFR) levels, or onset of end-stage renal disease or dialysis treatment, or kidney transplantation)after tonsillectomy

SECONDARY OUTCOMES:
Remission of proteinuria (complete or partial) | every 3-12months for 10 years after tonsillectomy
  The remission rate of proteinuria (include complete or partial remission )
Remission of hematuria (complete or partial) | every 3-12months for 10 years after tonsillectomy
  The remission rate of hematuria (include complete or partial remission )
Repeat renal biopsy | the fifth and tenth year after tonsillectomy
  reevaluate the renal histological changes by the Lee's glomerular grading
Side effects | every 3-12months for 10 years after tonsillectomy
  The shortterm and longterm side effects of tonsillectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363